CLINICAL TRIAL: NCT03768258
Title: Testosterone Implants and the Incidence of Breast Cancer RETROSPECTIVE CHART REVIEW
Brief Title: Testosterone Implants and the Incidence of Breast Cancer
Acronym: TIBCaP
Status: Completed | Type: Observational
Sponsor: Millennium Wellness LLC (Other)
Responsible Party: Principal Investigator, Rebecca L. Glaser, M.D., Physician, PI, Millennium Wellness LLC
Other Study IDs: MW0318-TBCP10Y
Record Dates: First submitted 2018-12-04; First posted 2018-12-07 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-08

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Testosterone; Anastrozole

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Testosterone Implant — Testosterone implants or combination testosterone + anstrozole implants used to treat symptoms of hormone/androgen deficiency
  Other Names: Testosterone + anastrozole implant

SUMMARY:
This current chart review study was designed to investigate the incidence of breast cancer in women treated with subcutaneous testosterone therapy for symptoms of hormone deficiency.

DETAILED DESCRIPTION:
A prior ten-year prospective, observational, study was initially approved in March of 2008 by the IRB board through the Atrium Medical Center, Premier Health Partners in Middletown, Ohio 45005 and registered through the Office for Human Research Protections (OHRP). Expedited approval continued annually through 2013 at which time the IRB board was closed. All participants signed a study consent and HIPPA consent. Recruitment closed in 2013. The original protocol was designed to investigate the incidence of breast cancer in women presenting with symptoms of hormone deficiency treated with subcutaneous testosterone implants or, testosterone combined with the aromatase inhibitor anastrozole implants. A computer program was specifically designed to track and follow patients prospectively and all patients continued to be followed through 2018.

ELIGIBILITY:
Inclusion Criteria:

* Female patients treated between March 2008 - March 2013
* Women who received at least two testosterone pellet insertion procedures
* Women previously accrued to the prospective cohort study

Exclusion Criteria:

* Pre-existing breast cancer
* Women who received a single testosterone pellet insertion

Ages: 24 Years to 92 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Women who presented to the office of Dr. Rebecca Glaser between March 2008- March of 2103 with symptoms of hormone deficiency and received testosterone implant therapy were asked to participate in the study. This current chart review study will examine the 10-year incidence of breast cancer in women accrued to the study.
Sampling Method: Probability Sample
Enrollment: 1268 (Actual)
Dates: Start 2008-03 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Incidence of invasive breast cancer | 10-year results
  The incidence of invasive breast cancer in women treated with testosterone therapy

SECONDARY OUTCOMES:
Incidence of ductal carcinoma in situ | 10-year results
  The incidence of DCIS in women treated with testosterone therapy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Glaser RL, York AE, Dimitrakakis C. Incidence of invasive breast cancer in women treated with testosterone implants: a prospective 10-year cohort study. BMC Cancer. 2019 Dec 30;19(1):1271. doi: 10.1186/s12885-019-6457-8. PMID 31888528
- See also: Statistical Methods and Results Additional File 1 — https://link.springer.com/article/10.1186/s12885-019-6457-8#Sec16